CLINICAL TRIAL: NCT01567826
Title: Reduction in YEllow Plaque by Aggressive Lipid LOWering Therapy. (YELLOW Trial)
Brief Title: Reduction in YEllow Plaque by Aggressive Lipid LOWering Therapy
Acronym: YELLOW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Annapoorna Kini (Other)
Responsible Party: Sponsor-Investigator, Annapoorna Kini, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 09-1294; IF1292822
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease
Keywords: YELLO; Atorvastatin; Simvastatin; Rosuvastatin; lipid therapy; Statin therapy; Coronary artery disease; CHD
MeSH Terms: conditions — Coronary Artery Disease | interventions — Simvastatin; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard of care lipid therapy (Active Comparator): standard-care lipid-lowering therapy: Zocor or Lipitor
  Interventions: Drug: standard of care lipid therapy
- aggressive lipid therapy (Experimental): aggressive lipid therapy: Crestor
  Interventions: Drug: Aggressive lipid therapy

INTERVENTIONS:
Drug: standard of care lipid therapy — Patients will be randomized in a 1:1 fashion to receive either A) Rosuvastatin (Crestor) 40mg daily, or B) standard-care lipid-lowering therapy.
  Zocor, Lipitor [any dose] and Crestor [less than 40mg]
  Other Names: Zocor; Lipitor; (Zocor, Lipitor, Crestor)
  Arms: standard of care lipid therapy
Drug: Aggressive lipid therapy — Patients will be randomized in a 1:1 fashion to receive either A) Rosuvastatin (Crestor) 40mg daily, or B) standard-care lipid-lowering therapy.
  Other Names: Rosuvastatin; Crestor
  Arms: aggressive lipid therapy

SUMMARY:
The study will assess the regression of yellow plaque content of the lipid pool after aggressive lipid therapy by utilizing NIR spectroscopy. Statin therapy using Rosuvastatin 10-40 mg will be compared to the statin therapy of either Atorvastatin or Simvastatin. This is a single site study. A total of 100 subjects will randomized, of which 40 will receive intensive lipid therapy (Rosuvastatin 40mg) and 40 will receive standard care lipid lowering therapy.

DETAILED DESCRIPTION:
Coronary artery disease (CHD) remains to be a leading cause of death in most countries (1) (2). It is well known that reducing cholesterol level by statin therapy is associated with significant reduction in plaque burden. REVERSAL (3) and ASTEROID (4) trials showed that in patients with coronary artery disease lipid-lowering with atorvastatin or rosuvastatin respectively reduced progression of coronary atherosclerosis and even cause repression of some lesions. CHD clinical events are related to plaque instability due to lipid content within the atherosclerotic plaque. High dose atorvastatin has shown to reduce the plaque lipid contents on serial IVUS analysis at 12 months. Therefore reduction in lipid content and thereby the plaque burden by lipid lowering therapy may stabilize the plaque and reduce cardiovascular events. High sensitivity C-reactive Protein (HsCRP) is an inflammatory biomarker that independently predicts future vascular events. In JUPITER (5) trial rosuvastatin (Crestor) significantly reduced the incidence of major cardiovascular events in apparently healthy people with elevated HsCRP. IVUS was utilized to demonstrate change in coronary artery vessel wall morphology over a relatively short period of time, but provided no data on the lipid content in the vessel wall. The application of NIR spectroscopy to identify lipid deposition within coronary arteries has been validated in ex vivo studies. Infrared spectra are collected as follows: Light of discrete wavelengths from a laser is directed onto the tissue sample via glass fibers. Light scattered from the samples is collected in fibers and launched into a spectrometer. The plot of signal intensity as a function of wavelength was used to develop chemometric models to discriminate lipid-cores from non-atherosclerotic tissue, and from atherosclerotic tissue that is predominantly fibrotic and from blood elements.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years of age and willing to participate
* Stable patients who will undergo cardiac catheterization and PCI (intent to stent)
* Patient is willing to go on a cholesterol lowering medication for the duration of the study and willing to change statin therapy to the randomized statin therapy regardless of previous statin therapy and dose (e.g. Atorvastatin 80 mg) Patients that are screened for this study and are receiving another Statin such as Pravachol will be required to be willing to change their therapy to Rosuvastatin as per is randomization. If patients are receiving another statin, such as pravachol, or any other agent, and are at appropriate Lipid levels, they will be permitted to continue this therapy (if randomized to the standard therapy arm). There are a virtually unlimited number of possible scenarios for potential combination of all Lipid lowering agents at the time of enrollment that patients may be taking.
* Signed written Informed Consent
* Women of childbearing potential must agree to be on an acceptable method of birth control/contraceptive such as barrier method (condoms/diaphragm); hormonal contraceptives (birth control pills, implants (Norplant) or injections (Depo-Provera)); Intrauterine Device; or abstinence (no sexual activity).
* Fluency in English and/or Spanish

Exclusion Criteria:

* Patients who have acute myocardial infarction (Q wave or non-Q wave with CK-MB > 5 times above the upper normal (31.5 ng/ml) within 72 hours)
* Patients who are in cardiogenic shock
* Patients with left main disease or restenotic lesions
* Patients with elevated CK-MB (> 6.5 ng/ml) or Tnl (> 0.5ng/L) at baseline
* Patients with platelet count < 100,000 cell/mm3
* Patients who have co-morbidity which reduces life expectancy to one year
* Patients who are currently participating in another investigational drug/device study
* Patients with known hypersensitivity to HMG CO-A reductase therapy (statins)
* Patients with liver disease
* Patient with creatinine > 2.0 mg/dL
* Pregnant women and women of childbearing potential who intend to have children during the duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna Kini, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Kini AS, Baber U, Kovacic JC, Limaye A, Ali ZA, Sweeny J, Maehara A, Mehran R, Dangas G, Mintz GS, Fuster V, Narula J, Sharma SK, Moreno PR. Changes in plaque lipid content after short-term intensive versus standard statin therapy: the YELLOW trial (reduction in yellow plaque by aggressive lipid-lowering therapy). J Am Coll Cardiol. 2013 Jul 2;62(1):21-9. doi: 10.1016/j.jacc.2013.03.058. Epub 2013 May 1. PMID 23644090
- [Derived] Dohi T, Maehara A, Moreno PR, Baber U, Kovacic JC, Limaye AM, Ali ZA, Sweeny JM, Mehran R, Dangas GD, Xu K, Sharma SK, Mintz GS, Kini AS. The relationship among extent of lipid-rich plaque, lesion characteristics, and plaque progression/regression in patients with coronary artery disease: a serial near-infrared spectroscopy and intravascular ultrasound study. Eur Heart J Cardiovasc Imaging. 2015 Jan;16(1):81-7. doi: 10.1093/ehjci/jeu169. Epub 2014 Sep 4. PMID 25190072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 779 patients consecutive patients with chronic stable angina presenting for elective coronary angiography were screened from May 21, 2010 until Jan 10, 2012. 87 participants met criteria and were randomized.
Groups:
- Standard of Care Lipid Therapy: standard-care lipid-lowering therapy: Zocor or Lipitor
  standard of care lipid therapy: Patients will be randomized in a 1:1 fashion to receive either A) Rosuvastatin (Crestor) 40mg daily, or B) standard-care lipid-lowering therapy.
  Zocor, Lipitor [any dose] and Crestor [less than 40mg]
Period: Overall Study
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Started | 43 | 44
Completed | 40 | 42
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.8) | 64.4 (9.29) | 63.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 31 | 35 | 66
Current tobacco use [Number; unit: participants]
  yes | 4 | 9 | 13
  no | 39 | 35 | 74
Hypertension [Number; unit: participants]
  yes | 40 | 40 | 80
  no | 3 | 4 | 7
Hypercholesterolemia [Number; unit: participants]
  yes | 40 | 39 | 79
  no | 3 | 5 | 8
Diabetes mellitus [Number; unit: participants] — (treated with insulin)
  participants
    yes | 3 | 5 | 8
    no | 40 | 39 | 79
Prior CVA/TIA [Number; unit: participants] — Cerebrovascular accident (CVA); Transient ischemic attack (TIA)
  participants
    yes | 3 | 2 | 5
    no | 40 | 42 | 82
Previous MI [Number; unit: participants] — Myocardial infarction (MI)
  participants
    yes | 8 | 8 | 16
    no | 35 | 36 | 71
Previous PCI [Number; unit: participants] — Percutaneous coronary intervention (PCI)
  participants
    yes | 20 | 16 | 36
    no | 23 | 28 | 51
Statin Use [Number; unit: participants]
  yes | 35 | 37 | 72
  no | 8 | 7 | 15
Beta-blocker use [Number; unit: participants]
  yes | 30 | 33 | 63
  no | 13 | 11 | 24
ACE-I/ARB use [Number; unit: participants] — Angiotensin-converting enzyme inhibitor (ACE-I); Angiotensin receptor blocker (ARB)
  participants
    yes | 19 | 16 | 35
    no | 24 | 28 | 52
Creatinine [Mean (Standard Deviation); unit: mg/dl] | 1.1 (1.3) | 1.0 (0.3) | 1.04 (0.96)
LAD Coronary vessel [Number; unit: participants] — Left anterior descending (LAD)
  participants
    yes | 17 | 20 | 37
    no | 26 | 24 | 50
LCx coronary vessel [Number; unit: participants] — Left circumflex (LCx)
  participants
    yes | 14 | 14 | 28
    no | 29 | 30 | 59
RCA coronary vessel [Number; unit: participants] — Right coronary artery (RCA)
  participants
    yes | 13 | 10 | 23
    no | 30 | 34 | 64

OUTCOME MEASURES:

1. Primary Outcome: Lipiscan - Lipid Core Burden Index (LCBI)
Description: The regression of yellow plaque content from the atherosclerotic lipid pool after statin therapy by utilizing NIR spectroscopy as compared from baseline to 6-8 weeks after intervention. Spectroscopic information obtained from raw spectra was transformed into a probability of lipid core that was mapped to a red-to-yellow color scale, with the low probability of lipid shown as red and the high probability of lipid shown as yellow. Analyses were performed offline using the Matlab-based software, as previously published. Yellow pixels within the analyzed segment were divided by all viable pixels to generate the lipid-core burden index (LCBI). The maximal value of LCBI for each nonculprit obstructive lesion was recorded and used for comparison.
Time Frame: at baseline and at 6-8 weeks after intervention
Population: Data were not available in 17 patients because of loss to follow-up (n = 5), incorrect image formatting that could not be recovered at the time of core laboratory analysis (n = 5), NIRS console/catheter malfunction at the time of index PCI (n = 3), and loss of disc integrity or corruption before core laboratory analysis (n = 4).
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Number analyzed (Participants) | 34 | 36
ratio
  Baseline LCBI, lesion | 95.4 [29.6 to 174.6] | 132.4 [99.0 to 201.2]
  Follow-up LCBI, lesion | 99.9 [38.2 to 204.3] | 99.8 [64.2 to 159.3]

2. Primary Outcome: LCBI4mm Max
Description: LCBI4mm max = change in lipid-core burden index at the 4-mm maximal segment. Spectroscopic information obtained from raw spectra was transformed into a probability of lipid core that was mapped to a red-to-yellow color scale, with the low probability of lipid shown as red and the high probability of lipid shown as yellow. Yellow pixels within the analyzed segment were divided by all viable pixels to generate the lipid-core burden index (LCBI). The maximal value of LCBI for each nonculprit obstructive lesion was recorded and used for comparison.
Time Frame: at baseline and at 6-8 weeks after intervention
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Number analyzed (Participants) | 34 | 36
ratio
  Baseline LCBI4mm max | 356.7 [145.2 to 509.2] | 490.6 [363.8 to 689.7]
  Follow-up LCBI4mm max | 385.7 [139.2 to 510.9] | 336.1 [252.3 to 479.9]

3. Primary Outcome: Change in LCBI4mm Max
Description: Change in LCBI4mm max at 6-8 weeks after intervention as compared to baseline. LCBI4mm max = change in lipid-core burden index at the 4-mm maximal segment.
Time Frame: at baseline and at 6-8 weeks after intervention
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: ratio
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Number analyzed (Participants) | 34 | 36
ratio | 2.4 [-36.1 to 44.7] | -149.1 [-210.9 to -42.9]
Statistical Analysis 1: Comparison: Standard of Care Lipid Therapy vs Aggressive Lipid Therapy; Test type: Superiority or Other; p = 0.01, ANCOVA

4. Primary Outcome: Change in LCBI, Lesion
Description: Change in LCBI at 6-8 weeks after intervention as compared to baseline
Time Frame: at baseline and at 6-8 weeks post intervention
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: ratio
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Number analyzed (Participants) | 34 | 36
ratio | 8.0 [-7.7 to 22.1] | -22.5 [-59.2 to -3.5]
Statistical Analysis 1: Comparison: Standard of Care Lipid Therapy vs Aggressive Lipid Therapy; Test type: Superiority or Other; p = 0.02, ANCOVA

5. Secondary Outcome: Intravascular Ultrasound (IVUS) Parameters
Description: Change in atheroma volume and lumen CSA on IVUS as related to change in yellow plaque index as compared from baseline to 6-8 weeks after intervention.
  Data not analyzed. Data not available.
Time Frame: at baseline and at 6-8 weeks after intervention
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Number analyzed (Participants) | 43 | 44
mm^2
  Baseline Total atheroma volume | 193.7 (61.7) | 195.8 (63.3)
  6-8 weeks Total atheroma volume | 199.6 (63.9) | 209.6 (74.1)
  Baseline Lumen CSA | 2.4 (0.6) | 2.5 (0.8)
  6-8 weeks Lumen CSA | 2.4 (0.7) | 2.5 (0.7)

6. Secondary Outcome: Fractional Flow Reserve (FFR) Value
Description: Change in FFR as related to change in yellow plaque index as compared from baseline to 6-8 weeks after intervention. Fractional flow reserve (FFR), defined as the ratio of maximum flow in the presence of a stenosis to normal maximum flow, is a lesion-specific index of stenosis severity that can be calculated by simultaneous measurement of mean arterial, distal coronary, and central venous pressure.
Time Frame: at baseline and at 6-8 weeks after intervention
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Number analyzed (Participants) | 43 | 44
ratio
  Baseline | 0.73 (0.1) | 0.73 (0.1)
  Follow-up | 0.73 (0.1) | 0.75 (.01)

7. Secondary Outcome: Diameter Stenosis
Description: Percentage stenosis of vessel diameter in the analysis segment of nontarget lesions as measured by angiography that remained >70%, after successful PCI of the target lesion.
Time Frame: Baseline and 6-8 weeks post intervention
Measure: Number; unit: percentage of lesions
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Number analyzed (Participants) | 43 | 44
percentage of lesions
  Baseline | 79.9 | 79.6
  Follow-up | 83 | 79.4

8. Secondary Outcome: Post PCI Cardiac Enzymes
Description: Correlation of yellow plaque index with post procedure CK-MB, Troponin-I release.
Time Frame: at 6-8 weeks after intervention
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Number analyzed (Participants) | 43 | 44
ng/mL
  CK-MB | 5.1 (9.0) | 3.7 (0.3)
  Troponin-I | 0.4 (1.0) | 0.3 (5.1)

9. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: MACE defined as a combined clinical endpoint of death, MI (Q wave or non Q-wave with CK-MB >3 times above the upper normal limit (48 U/L), urgent revascularization or stroke at 30 days and 1 year. Details reported in adverse events section.
Time Frame: at 6-8 weeks after intervention
Measure: Number; unit: participants
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Number analyzed (Participants) | 43 | 44
participants | 2 | 3

10. Secondary Outcome: Blood Chemistry - HsCRP
Description: Correlation of yellow plaque index with changes in levels of blood HsCRP as compared from baseline to 6-8 weeks after intervention
Time Frame: at baseline and at 6-8 weeks after intervention
Measure: Median (Inter-Quartile Range); unit: mg/l
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Number analyzed (Participants) | 43 | 44
mg/l
  Baseline | 1.7 [0.7 to 3.4] | 1.7 [0.8 to 3.5]
  Follow-Up | 1.9 [0.7 to 4.7] | 1.2 [0.7 to 2.5]

ADVERSE EVENTS:
Arm/Group | Standard of Care Lipid Therapy | Aggressive Lipid Therapy
Serious Adverse Events (participants affected / at risk) | 2/43 | 3/44
Other Adverse Events (participants affected / at risk) | 9/43 | 7/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care Lipid Therapy (N=43) | Aggressive Lipid Therapy (N=44)
Hospitalization (Cardiac disorders) | 2 | 3 — Hospitalization for Chest Pain
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Lipid Therapy (N=43) | Aggressive Lipid Therapy (N=44)
Unplanned revascularization (Vascular disorders) | 2 (2) | 0 (0)
Periprocedural complications (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Any bleeding (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
AST > 3x ULN (Hepatobiliary disorders) | 0 (0) | 0 (0) — aspartate aminotransferase (AST); upper limit of normal (ULN)
ALT > 3x ULN (Hepatobiliary disorders) | 0 (0) | 0 (0) — alanine aminotransferase (ALT); upper limit of normal (ULN)
Creatine kinase-MB > 5x ULN (Renal and urinary disorders) | 2 (2) | 1 (1)
Creatine kinase-MB >10x ULN (Renal and urinary disorders) | 2 (2) | 0 (0)
Statin discontinuation (General disorders) | 0 (0) | 0 (0)
Statin dose reduction (General disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Limitations - small sample size and short duration of follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes